CLINICAL TRIAL: NCT01193439
Title: Safety of Thoracoscopy in Patients With High Risk
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Muzaffer Metintas, MD, Eskisehir Osmangazi University
Other Study IDs: 082010/1
Record Dates: First submitted 2010-08-26; First posted 2010-09-02 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Pleural Diseases
Keywords: thoracoscopy; pleural diseases; complications; safety
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with high risk
- Patients in normal conditions

SUMMARY:
Medical thoracoscopy can be performed for diagnostic as well as therapeutic purposes. Thoracoscopy in the diagnosis of pleural diseases is highly sensitive for detecting pleural neoplasia with negative pleural fluid cytology and in the diagnosis of tuberculosis. The indication of thoracoscopy in patients with pleural effusion has been optimized. In some studies medical thoracoscopy has been claimed a useful diagnostic tool with a very low rate of complications. However the investigators do not know its safety on high risk patients. Because many patients having suspected malignancy have bed conditions due to other health problems such as coronary heart diseases, COPD, arrythmia, hypoxemia. In this study the investigators aimed to test the safety of medical thoracoscopy in the patients with high risk for complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with exudative pleural effusion

Exclusion Criteria:

* Patients without pleural effusion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require thoracoscpic investigation
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2002-01; Primary Completion 2009-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 years
  All participants will have been followed for side effects of medical thoracoscopy. All side effects established in the special forms designed for this study. Side effects measured and recorded according to each characteristic such as pain, air leakege, pneumothorax, empyema, local infection, haemorragy etc.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Metintas, Professor, Principal Investigator — Head of Department, Professor of pulmonary medicine
Locations (1):
- ESOGU, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Rodriguez-Panadero F. Medical thoracoscopy. Respiration. 2008;76(4):363-72. doi: 10.1159/000158545. Epub 2008 Nov 12. PMID 19018161